CLINICAL TRIAL: NCT00606476
Title: A Phase II, Multicenter, Open-Label, Long-Term Treatment Study to Determine the Safety, Tolerability, and Efficacy of Bapineuzumab (AAB-001) in Patients With Alzheimer's Disease Who Participated in Study AAB-001-201 or AAB-001-102
Brief Title: AAB-001 (Bapineuzumab) Open-Label, Long-Term Extension Study in Patients With Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AAB-001-251
Record Dates: First submitted 2008-01-11; First posted 2008-02-04 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2012-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 0.15 mg/kg active bapineuzumab
  Interventions: Drug: Bapineuzumab (AAB-001)
- 2 (Active Comparator): 0.5 mg/kg active bapineuzumab
  Interventions: Drug: Bapineuzumab (AAB-001)
- 3 (Active Comparator): 1.0 mg/kg active bapineuzmab
  Interventions: Drug: Bapineuzumab (AAB-001)

INTERVENTIONS:
Drug: Bapineuzumab (AAB-001) — IV q13w
  Other Names: AAB-001

SUMMARY:
This is a multicenter, open-label, long-term extension study in male and female patients with mild to moderate Alzheimer's Disease (AD) who must have completed one of the following studies: AAB-001-201 or AAB-001-102. All patients enrolled in Study AAB-001-251 will receive infusions of AAB-001 (bapineuzumab), including patients randomized to placebo in Study 201 and 102. Approximately 30 study sites in the US will be involved. Each patient's participation may vary from 3 months up to 84 months depending on the date of enrollment in this study.

AAB-001 (bapineuzumab) is a humanized monoclonal antibody, which binds to and potentially clears beta amyloid peptide, and is designed to provide antibodies to beta amyloid directly to the patient.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet ALL of the following criteria to be considered for enrollment into this study:

1. Signed and dated written informed consent obtained from the subject and/or the subject's caregiver in accordance with the local regulations.
2. Subjects must have completed Study 201 Visit 22 (Week 78), or Study 102 Visit 11 (Week 16).
3. Magnetic resonance imaging scan of sufficient quality for the Radiologist to evaluate subject safety from Study 201 Visit 21 (Week 71), or Study 251 Screening Visit for subjects from Study 102.
4. Lives at home with appropriate caregiver capable of accompanying the subject on all clinic visits, or community dwelling with caregiver capable of accompanying the subject on all clinic visits and visiting with the subject approximately five times per week for the duration of the study.
5. In the opinion of the investigator, the subject and the caregiver will be compliant.

Exclusion Criteria:

ANY one of the following will exclude a subject from being enrolled into the study:

1. Significant neurological disease other than AD that may affect cognition.
2. Screening visit brain MRI scan (ie, Study 201 Visit 21 (Week 71), or for Study 102, the Study 251 Screening Visit) indicative of any other significant abnormality including but not limited to multiple microhemorrhages or evidence of a single prior hemorrhage >1 cm3, multiple lacunar infarcts or evidence of a single prior infarct >1 cm3, evidence of a cerebral contusion, encephalomalacia, arachnoid cysts, or brain tumors (eg, meningioma) unless approved by the medical monitor.
3. Current presence of a clinically significant major psychiatric disorder according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV) or any clinically significant symptom that could affect the subject's ability to participate in the study.
4. Current clinically significant systemic illness that is likely to result in deterioration of the subject's condition or affect the subject's safety during the study.
5. History of clinically evident stroke or history of clinically significant carotid or vertebrobasilar stenosis or plaque.
6. History of seizures, excluding febrile seizures in childhood.
7. Weight greater than 120 kg (264 lbs).
8. History or evidence of any clinically significant autoimmune disease or disorder of the immune system.
9. Clinically significant infection within the last 30 days (eg, chronic persistent or acute infection).
10. Treatment with immunosuppressive medications (eg, systemic corticosteroids) within the last 90 days (topical and nasal corticosteroids and inhaled corticosteroids for asthma are permitted) or chemotherapeutic agents for malignancy within the last three years.
11. Myocardial infarction within the last two years.
12. History of cancer within the last five years, with the exception of basal cell carcinoma, and nonmetastatic squamous cell carcinoma of the skin.
13. Other clinically significant abnormality on screening (ie, Study 201 Visit 22 [Week 78], or Study 102 Visit 11 [Week 16]) physical, neurological, laboratory, or ECG examination (eg, atrial fibrillation) that could compromise the study or be detrimental to the subject.
14. Hemoglobin less than 11 g/dL at screening (ie, Study 201 Visit 22 [Week 78], or Study 102 Visit 11 [Week16]).
15. Smoking more than 20 cigarettes per day.
16. History of alcohol or drug dependence or abuse within the last two years.
17. Current use of anticonvulsant for seizures, anti-Parkinson's, anticoagulant (excluding the use of aspirin 325 mg/day or less), or narcotic medications.
18. Any prior experimental treatment with AN1792 or other experimental immunotherapeutic or vaccine for AD (other than bapineuzumab).
19. Any known hypersensitivity to any of the excipients contained in the study drug formulation.
20. Women of childbearing potential.
21. Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, cerebrospinal fluid (CSF) shunts, metal fragments or foreign objects in the eyes, skin, or body that would contraindicate a brain MRI scan (unless otherwise approved by the Sponsor and/or its designees).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2006-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of long-term treatment of bapineuzumab in subjects with AD. | 3-84 months
  * The incidence and severity of treatment-emergent adverse events (TEAEs);
  * Clinically important changes in safety assessment results (including, as appropriate, vital signs, weight, clinical laboratory tests, electrocardiograms [ECGs], brain magnetic resonance imaging [MRIs], physical and neurological examinations, and infusion site assessments).

SECONDARY OUTCOMES:
To evaluate the efficacy of long-term treatment of bapineuzumab in subjects with AD. | 3-84 months
  Change from Visit 2 (Pre-Day 1) and Visit 22 (Week 78) of Study AAB-001-201 for the following scales:
  * Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-Cog)
  * Disability Assessment for Dementia (DAD)
  * Mini Mental State Examination (MMSE)
  Change from Study AAB-001-251Visit 1 (Day 1) for the following scales:
  * Dependence Scale
  * Resource Utilization in Dementia (RUD) Lite
  Change from Study 251 Screening Visit for the following scales for subjects entering from Study AAB-001-102 (US):
  * ADAS-Cog
  * DAD
  * MMSE

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Janssen AI Investigational Site, Peoria, Arizona
  - Janssen AI Investigational Site, Sun City, Arizona
  - Janssen AI Investigational Site, Encino, California
  - Janssen AI Investigational Site, Irvine, California
  - Janssen AI Investigational Site, La Jolla, California
  - Janssen AI Investigational Site, Los Alamitos, California
  - Janssen AI Investigational Site, Sacramento, California
  - Janssen AI Investigational Site, San Francisco, California
  - Janssen AI Investigational Site, New Haven, Connecticut
  - Janssen AI Investigational Site, Washington D.C., District of Columbia
  - Janssen AI Investigational Site, Delray Beach, Florida
  - Janssen AI Investigational Site, Jacksonville, Florida
  - Janssen AI Investigational Site, Chicago, Illinois
  - Janssen AI Investigational Site, Indianapolis, Indiana
  - Janssen AI Investigational Site, Boston, Massachusetts
  - Janssen AI Investigational Site, Ann Arbor, Michigan
  - Janssen AI Investigational Site, Rochester, Minnesota
  - Janssen AI Investigational Site, St Louis, Missouri
  - Janssen AI Investigational Site, Eatontown, New Jersey
  - Janssen AI Investigational Site, New York, New York
  - Janssen AI Investigational Site, Rochester, New York
  - Janssen AI Investigational Site, Durham, North Carolina
  - Janssen AI Investigational Site, Portland, Oregon
  - Janssen AI Investigational Site, Pittsburgh, Pennsylvania
  - Janssen AI Investigational Site, Providence, Rhode Island
  - Janssen AI Investigational Site, Dallas, Texas
  - Janssen AI Investigational Site, Houstan, Texas
  - Janssen AI Investigational Site, Bennington, Vermont
  - Janssen AI Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Salloway S, Marshall GA, Lu M, Brashear HR. Long-Term Safety and Efficacy of Bapineuzumab in Patients with Mild-to-Moderate Alzheimer's Disease: A Phase 2, Open-Label Extension Study. Curr Alzheimer Res. 2018;15(13):1231-1243. doi: 10.2174/1567205015666180821114813. PMID 30129411
- [Derived] Arrighi HM, Barakos J, Barkhof F, Tampieri D, Jack C Jr, Melancon D, Morris K, Ketter N, Liu E, Brashear HR. Amyloid-related imaging abnormalities-haemosiderin (ARIA-H) in patients with Alzheimer's disease treated with bapineuzumab: a historical, prospective secondary analysis. J Neurol Neurosurg Psychiatry. 2016 Jan;87(1):106-12. doi: 10.1136/jnnp-2014-309493. Epub 2015 Feb 10. PMID 25669746